CLINICAL TRIAL: NCT01844531
Title: Bioequivalence of Empagliflozin/Metformin (500 mg) Fixed Dose Combination Tablets Compared to Single Tablets Administered Together in Healthy Male and Female Volunteers Under Fed Conditions (an Open-label, Randomised, Single-dose, Four-way Crossover Study)
Brief Title: Bioequivalence of Empagliflozin and Metformin Given as a Fixed Dose Combination Compared to Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.6; 2012-000082-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (4):
- FDC empagliflozin dose 1 and metformin (Experimental): fix dose combination tablet after intake of a high fat, high caloric meal
  Interventions: Drug: empagliflozin and metformin
- empagliflozin dose 1 + metformin tablets (Active Comparator): single tablets after intake of a high fat, high caloric meal
  Interventions: Drug: empagliflozin; Drug: metformin (Glucophage®)
- FDC empagliflozin dose 2 and metformin (Experimental): fix dose combination tablet after intake of a high fat, high caloric meal
  Interventions: Drug: empagliflozin and metformin
- empagliflozin dose 2 + metformin tablets (Active Comparator): single tablets after intake of a high fat, high caloric meal
  Interventions: Drug: metformin (Glucophage®); Drug: empagliflozin

INTERVENTIONS:
Drug: empagliflozin — single tablet empagliflozin
  Arms: empagliflozin dose 1 + metformin tablets
Drug: metformin (Glucophage®) — single tablet metformin
  Arms: empagliflozin dose 1 + metformin tablets
Drug: metformin (Glucophage®) — single tablet metformin
  Arms: empagliflozin dose 2 + metformin tablets
Drug: empagliflozin — single tablet empagliflozin
  Arms: empagliflozin dose 2 + metformin tablets
Drug: empagliflozin and metformin — FDC tablet empagliflozin and metformin
  Arms: FDC empagliflozin dose 1 and metformin
Drug: empagliflozin and metformin — FDC tablet empagliflozin and metformin
  Arms: FDC empagliflozin dose 2 and metformin

SUMMARY:
The primary objective of this trial is to establish bioequivalence of two fixed dose combination (FDC) tablets (containing medium dose empagliflozin/500 mg metformin [Test 1] and low dose empagliflozin/500 mg metformin [Test 2]) and of the single tablets (medium dose empagliflozin tablets + Glucophage® 500 mg tablet [Reference 1] and low dose empagliflozin tablet + Glucophage® 500 mg tablet [Reference 2]) when administered together after a high fat, high caloric meal.

The assessment of safety and tolerability will be an additional objective of this trial.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects
2. Subjects must be able to understand and comply with study requirements
3. Age 18 to 50 years
4. Body mass index (BMI) 18.5 to 29.9 kg/m2

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.6.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- FDC Empa12.5/ Empa12.5+Met500/ FDC Empa5/ Empa5+Met500: Participants first received Treatment T1 (12.5 mg empagliflozin/500 mg metformin Fixed Dose Combination (FDC)). After a washout phase of at least 5 days, they then received Treatment R1 (12.5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T2 (5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R2 (5 mg empagliflozin and 500 mg metformin, single tablets). Oral administration.
- Empa12.5+Met500/ FDC Empa12.5/ Empa5+Met500/ FDC Empa5: Participants first received Treatment R1 (12.5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T1 (12.5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R2 (5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T2 (5 mg empagliflozin/500 mg metformin FDC). Oral administration.
- FDC Empa5/ Empa5+Met500/ FDC Empa12.5/ Empa12.5+Met500: Participants first received Treatment T2 (5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R2 (5 mg empagliflozin and 500 mg metformin, single tablets)Treatment T1 (12.5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R1 (12.5 mg empagliflozin and 500 mg metformin, single tablets). Oral administration.
- Empa5+Met500/ FDC Empa5/ Empa12.5+Met500/ FDC Empa12.5: Participants first received Treatment R2 (5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T2 (5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R1 (12.5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T1 (12.5 mg empagliflozin/500 mg metformin FDC). Oral administration.
Period: Overall Study
Arm/Group | FDC Empa12.5/ Empa12.5+Met500/ FDC Empa5/ Empa5+Met500 | Empa12.5+Met500/ FDC Empa12.5/ Empa5+Met500/ FDC Empa5 | FDC Empa5/ Empa5+Met500/ FDC Empa12.5/ Empa12.5+Met500 | Empa5+Met500/ FDC Empa5/ Empa12.5+Met500/ FDC Empa12.5
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set, included all subjects that entered the study and had taken at least 1 dose of trial medication.
Groups:
- FDC Empa12.5/ Empa12.5+Met500/ FDC Empa5/ Empa5+Met500: Participants first received Treatment T1 (12.5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R1 (12.5 mg empagliflozin and 500 mg metformin, single tablets). After a washout phase of at least 5 days, they then received Treatment T2 (5 mg empagliflozin/500 mg metformin FDC). After a washout phase of at least 5 days, they then received Treatment R2 (5 mg empagliflozin and 500 mg metformin, single tablets).
  Oral administration.
- Total: Total of all reporting groups
Arm/Group | FDC Empa12.5/ Empa12.5+Met500/ FDC Empa5/ Empa5+Met500 | Empa12.5+Met500/ FDC Empa12.5/ Empa5+Met500/ FDC Empa5 | FDC Empa5/ Empa5+Met500/ FDC Empa12.5/ Empa12.5+Met500 | Empa5+Met500/ FDC Empa5/ Empa12.5+Met500/ FDC Empa12.5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (8.6) | 30.8 (7.6) | 35.8 (10.5) | 37.5 (9.0) | 35.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 4 | 15
  Male | 1 | 4 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞ for Empagliflozin
Description: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Empagliflozin
Time Frame: 1hour (h) before drug intake and 20minutes (min),40min,1h,1h 30min,2h,2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h,10h,12h,24h,34h,48h,72h after drug intake
Population: Pharmacokinetics set (PKS) included all treated subjects with at least 1 evaluable observation for at least 1 primary pharmacokinetic endpoint without important protocol violations relevant to the statistical evaluation of pharmacokinetics who had not taken any restricted medication and had not experienced emesis before or at 2 times median tmax
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- 12.5 mg Empagliflozin and 500 mg Metformin as FDC: 12.5 mg empagliflozin/500 mg metformin as Fixed Dose Combination, oral administration
- 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets: 12.5 mg empagliflozin and 500 mg metformin as single tablets, oral administration
- 5 mg Empagliflozin and 500 mg Metformin as FDC: 5 mg empagliflozin/500 mg metformin as Fixed Dose Combination, oral administration
- 5 mg Empagliflozin and 500 mg Metformin as Single Tablets: 5 mg empagliflozin and 500 mg metformin as single tablets, oral administration
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
nmol*h/L | 2780 (16.1) | 2870 (17.3) | 1110 (15.7) | 1070 (19.2)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUCinfpred [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA). The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale; Test type: Superiority or Other; p = 0.0000, ANOVA — Model included effects:sequence;subjects within sequences;period and treatment with subjects within sequences as random effect; Adjusted gMean ratio FDC/single tablets = 97.92, 90% CI 2-sided [93.529 to 102.520], Standard Error of Mean 8.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUCinfpred [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA). The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale; Test type: Superiority or Other; p < .0001, ANOVA — Model included effects:sequence;subjects within sequences;period and treatment with all effects as fixed; Adjusted gMean ratio FDC/single tablets = 98.00, 90% CI 2-sided [93.57 to 102.65], Standard Error of Mean 8.3 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500 , PK set AUCinfpred [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA). The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale; Test type: Superiority or Other; p = 0.0000, ANOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted gMean ratio FDC/single tablets = 102.79, 90% CI 2-sided [99.077 to 106.633], Standard Error of Mean 6.7 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 (T2) : Empa5 + Met500 (R2), PK set AUCinfpred [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 102.50, 90% CI 2-sided [98.78 to 106.36], Standard Error of Mean 6.7 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

2. Primary Outcome: AUC0-∞ for Metformin
Description: AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Metformin
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
ng*h/mL | 5590 (19.0) | 5820 (21.8) | 5960 (18.0) | 6190 (19.5)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUCinfpred [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0006, ANOVA; Adjusted gMean ratio FDC/single tablets = 96.25, 90% CI 2-sided [88.542 to 104.628], Standard Error of Mean 15.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 (T1) : Empa12.5 + Met500 (R1), PK set AUCinfpred [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0004, ANOVA; Adjusted gMean ratio FDC/single tablets = 97.21, 90% CI 2-sided [89.41 to 105.68], Standard Error of Mean 15.1 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500, PK set AUCinfpred [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 96.79, 90% CI 2-sided [91.772 to 102.093], Standard Error of Mean 9.8 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 : Empa5 + Met500, PK set AUCinfpred [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 96.91, 90% CI 2-sided [91.79 to 102.32], Standard Error of Mean 9.8 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

3. Secondary Outcome: AUC0-tz for Empagliflozin
Description: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) for Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
nmol*h/L | 2740 (16.3) | 2830 (17.3) | 1080 (15.7) | 1040 (19.1)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUClast [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 98.00, 90% CI 2-sided [93.530 to 102.686], Standard Error of Mean 8.5 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUClast [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 98.07, 90% CI 2-sided [93.55 to 102.81], Standard Error of Mean 8.5 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500, PK set AUClast [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 102.77, 90% CI 2-sided [99.146 to 106.522], Standard Error of Mean 6.5 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 : Empa5 + Met500, PK set AUClast [nmol*h/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 102.49, 90% CI 2-sided [98.85 to 106.25], Standard Error of Mean 6.5 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

4. Primary Outcome: Cmax for Empagliflozin
Description: Cmax (maximum measured concentration of the analyte in plasma) for Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
nmol/L | 294 (23.7) | 282 (27.4) | 109 (22.8) | 106 (22.5)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set Cmax [nmol/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 104.61, 90% CI 2-sided [99.882 to 109.555], Standard Error of Mean 8.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 : Empa12.5 + Met500, PK set Cmax [nmol/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 104.53, 90% CI 2-sided [99.76 to 109.53], Standard Error of Mean 8.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500, PK set Cmax [nmol/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 102.96, 90% CI 2-sided [97.917 to 108.258], Standard Error of Mean 9.2 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 : Empa5 + Met500, PK set Cmax [nmol/L] for EMPAGLIFLOZIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 102.80, 90% CI 2-sided [97.72 to 108.14], Standard Error of Mean 9.2 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

5. Primary Outcome: Cmax for Metformin
Description: Cmax (maximum measured concentration of the analyte in plasma) for Metformin
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
ng/mL | 686 (14.1) | 718 (19.7) | 693 (12.8) | 743 (19.6)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set Cmax [ng/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 94.76, 90% CI 2-sided [89.056 to 100.819], Standard Error of Mean 11.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 : Empa12.5 + Met500, PK set Cmax [ng/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 94.40, 90% CI 2-sided [88.64 to 100.54], Standard Error of Mean 11.4 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500, PK set Cmax [ng/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0002, ANOVA; Adjusted gMean ratio FDC/single tablets = 93.83, 90% CI 2-sided [88.006 to 100.034], Standard Error of Mean 11.9 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 : Empa5 + Met500, PK set Cmax [ng/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0003, ANOVA; Adjusted gMean ratio FDC/single tablets = 93.98, 90% CI 2-sided [87.94 to 100.43], Standard Error of Mean 12.0 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

6. Secondary Outcome: AUC0-tz for Metformin
Description: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) for Metformin
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Number analyzed (Participants) | 21 | 23 | 23 | 20
ng*h/mL | 5480 (18.9) | 5720 (21.2) | 5820 (17.7) | 6110 (19.2)
Statistical Analysis 1: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUClast [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0008, ANOVA; Adjusted gMean ratio FDC/single tablets = 95.78, 90% CI 2-sided [88.000 to 104.256], Standard Error of Mean 15.7 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: 12.5 mg Empagliflozin and 500 mg Metformin as FDC vs 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa12.5 : Empa12.5 + Met500, PK set AUClast [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0006, ANOVA; Adjusted gMean ratio FDC/single tablets = 96.74, 90% CI 2-sided [88.78 to 105.41], Standard Error of Mean 15.5 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 3: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability comparison FDC Empa5 : Empa5 + Met500, PK set AUClast [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p = 0.0000, ANOVA; Adjusted gMean ratio FDC/single tablets = 95.94, 90% CI 2-sided [91.199 to 100.934], Standard Error of Mean 9.3 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]
Statistical Analysis 4: Comparison: 5 mg Empagliflozin and 500 mg Metformin as FDC vs 5 mg Empagliflozin and 500 mg Metformin as Single Tablets; Adjusted by-treatment geometric means and relative bioavailability - analysis with fixed effects for all terms comparison FDC Empa5 : Empa5 + Met500, PK set AUClast [ng*h/mL] for METFORMIN (PLASMA EDTA); Test type: Superiority or Other; p < .0001, ANOVA; Adjusted gMean ratio FDC/single tablets = 96.10, 90% CI 2-sided [91.28 to 101.19], Standard Error of Mean 9.3 — *Results reported as Standard Error of the mean are Intra-individual geometric coefficient of variation [%]

ADVERSE EVENTS:
Time Frame: From study drug administration of 1 treatment period until study drug administration in the next treatment period or date of trial completion plus 1 day, up to 8 days (and up to 16 days for one subject only)
Arm/Group | 12.5 mg Empagliflozin and 500 mg Metformin as FDC | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets | 5 mg Empagliflozin and 500 mg Metformin as FDC | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 3/21 | 6/23 | 3/23 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12.5 mg Empagliflozin and 500 mg Metformin as FDC (N=21) | 12.5 mg Empagliflozin and 500 mg Metformin as Single Tablets (N=23) | 5 mg Empagliflozin and 500 mg Metformin as FDC (N=23) | 5 mg Empagliflozin and 500 mg Metformin as Single Tablets (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No